CLINICAL TRIAL: NCT01136590
Title: Multicenter, Randomized Placebo-controlled Clinical Trial to Evaluate the Effect of Perioperative Use of Tranexamic Acid on Transfusion Requirements and Surgical Bleeding in Major Spine Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Hospital Vall d'Hebron (Other); Hospital Clinic of Barcelona (Other); Hospital Universitari de Bellvitge (Other); Hospital Universitario Getafe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRANEX2009; 2008-006938-94 (EudraCT Number)
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Spinal Fusion; Antifibrinolytic Agents; Hemorrhage; Blood Transfusion
Keywords: Spinal deformity correction; Surgical bleeding; Transfusion practice; Spinal Fusion; Antifibrinolytic Agents; Hemorrhage; Blood Transfusion
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- tranexamic acid (Experimental): tranexamic acid will be administered as a bolus (10-mg/kg dose ) or as a fast, 20-minute intravenous infusion before performing the incision at the start of surgery, followed by perfusion of 2 mg/kg/hour up to the time the surgical wound is closed at completion of surgery
  Interventions: Drug: Tranexamic Acid
- placebo (Placebo Comparator): The placebo will be administered according to the same regimen and infusion time as the medication in the study arm (bolus or 20-minute fast infusion before the incision at the beginning of surgery followed by perfusion of 2 mg/kg/hour until closure of the surgical wound at completion of surgery)
  Interventions: Drug: fisiologic serum

INTERVENTIONS:
Drug: Tranexamic Acid — A 10-mg/kg dose of tranexamic acid will be administered as a bolus or as a fast, 20-minute intravenous infusion before performing the incision at the start of surgery, followed by perfusion of 2 mg/kg/hour up to the time the surgical wound is closed at completion of surgery.
  Arms: tranexamic acid
Drug: fisiologic serum — The placebo will be administered according to the same regimen and infusion time as the medication in the study arm (bolus or 20-minute fast infusion before the incision at the beginning of surgery followed by perfusion of 2 mg/kg/hour until closure of the surgical wound at completion of surgery)
  Arms: placebo

SUMMARY:
Current evidence regarding the efficacy and safety of perioperative administration of tranexamic acid for antifibrinolysis does not suffice to support its use in major spinal surgery.

OBJECTIVES: To evaluate the effectiveness of tranexamic acid for decreasing transfusion requirements and bleeding in this patient population. To evaluate the safety of this antifibrinolytic agent in the intraoperative and mid-term postoperative period.

METHODS: Multicenter, randomized, double-blind, placebo-controlled clinical trial with parallel groups. The main outcome measure is intraoperative and postoperative transfusion requirements; blood loss and safety will also be evaluated. Previous results in other types of surgery suggest that tranexamic acid reduces transfusion requirements and blood loss. Hence, the hypothesis of this study is that tranexamic acid will significantly reduce blood loss in comparison to a placebo in major spine surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old of both sexes
* scheduled for complex spine surgery
* ASA I-III
* weighing more than 30 kg
* body mass index <30 kg/m2
* operated on in the participating hospitals
* major spinal surgery
* signed an informed consent form to be included in the study

Exclusion Criteria:

* a history of allergy or hypersensitivity to the agent used
* receiving medication that can interfere with coagulation (acetylsalicylic acid, oral anticoagulants, or antiplatelet agents)
* a history of frequent bleeding
* plasma creatinine values >1.5 mg/dL in the baseline analysis
* platelet count less than 150,000/mm3 in the follow-up analysis
* abnormal prothrombin time (INR >1.5) or partial thromboplastin time (INR >1.5)
* a history of a thromboembolic episode before surgery
* family history of thromboembolism
* lack of consent to participate in the study
* infectious disease, tumor or trauma of the spine as the reason for surgery
* scheduled for surgery with an anterior and posterior surgical approach, whether sequential or on the same day

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2010-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the number of transfused units required during the intraoperative and postoperative period | 7 days postoperative period

SECONDARY OUTCOMES:
Total blood loss: intraoperative and postoperative values | 48 hours postoperative
  Intraoperative blood loss is evaluated by measuring the volume of suction aspirate and weighing the swabs with a precision digital scale. Postoperative blood loss is determined by recording the volume of blood collected through the suction drains at 24 and 48 hours.
Adverse events in the perioperative period, immediate postoperative period, and at mid-term | up to 6 weeks after the procedure
  Adverse events in the perioperative period, immediate postoperative period, and at mid-term (up to 6 weeks after the procedure) will be recorded, with special emphasis on follow-up of thrombotic events and clinically suspected deep venous thrombosis, renal function, and visual abnormalities reported by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Maria J Colomina, MD Ph, Study Chair — Hospital Vall d'Hebron; Misericordia Basora, MD Ph, Principal Investigator — Hospital Clinic of Barcelona; Maylin Koo, MD Ph, Principal Investigator — Hospital Universitari de Bellvitge; Javier Pizones, MD, Principal Investigator — Hospital de Getafe.
Locations (4):
- Spain (4):
  - Hospital Clinic de Barcelona, Barcelona, Barcelona
  - Hospital Vall d'Hebron de Barcelona, Barcelona, Barcelona
  - Hospital de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital de Getafe, Getafe, Madrid

REFERENCES:
- [Derived] Colomina MJ, Koo M, Basora M, Pizones J, Mora L, Bago J. Intraoperative tranexamic acid use in major spine surgery in adults: a multicentre, randomized, placebo-controlled trialdagger. Br J Anaesth. 2017 Mar 1;118(3):380-390. doi: 10.1093/bja/aew434. PMID 28203735